CLINICAL TRIAL: NCT02600052
Title: Efficacy of Pattern Respiratory Proprioceptive Neuromuscular Facilitation Associated With Aerobic Training on the Volumes, Lung Capacity and Six-minute Walking Test in Individuals With Parkinson: Randomized Clinical Trial
Brief Title: Efficacy of Pattern Respiratory PNF Associated Aerobic Training on Lung Volumes and 6MWT Test in Parkinson Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Carlos Rego Barros, researcher master, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06704028420
Record Dates: First submitted 2015-11-03; First posted 2015-11-09 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GPNF (Experimental): Patients will be submitted to aerobic training, with prior application of PNF technique and after its completion. Aerobic training program will consist of walking on a treadmill for 30 minutes with 5 minute initial heating and 5-minute cool-down. The training intensity will correspond to 60% of maximal oxygen consumption (VO2max) or 70% of maximum heart rate (MHR) predicted by age is determined by the formula: HR max = 208 - (0.7 x age). The speed and incline of the treadmill will be adjusted according to the patient's performance, so that they maintain the same intensity throughout the course of the training.
  Interventions: Other: PNF; Device: treadmill
- GCONTROL (Active Comparator): Patients will be submitted to aerobic training, with prior application of relax technique and after its completion. Aerobic training program will consist of walking on a treadmill for 30 minutes with 5 minute initial heating and 5-minute cool-down. The training intensity will correspond to 60% of maximal oxygen consumption (VO2max) or 70% of maximum heart rate (MHR) predicted by age is determined by the formula: HR max = 208 - (0.7 x age). The speed and incline of the treadmill will be adjusted according to the patient's performance, so that they maintain the same intensity throughout the course of the training.
  Interventions: Device: treadmill

INTERVENTIONS:
Other: PNF — RESPIRATORY PATTERN PROPRIOCEPTIVE NEUROMUSCULAR FACILITATION
  Arms: GPNF
Device: treadmill — AEROBIC TRAINING

SUMMARY:
INTRODUCTION:

Parkinson's disease (PD) is a neurodegenerative disorder that causes motor disorders such as bradykinesia, rigidity and tremor. In addition to the motor symptoms occurring in the overall PD patients, mostly there is associated respiratory disorders. The respiratory impairment may be due by postural changes, limiting the flexibility and expandability of the chest wall causing decreased lung volumes and flows. So the exercise Proprioceptive Neuromuscular Facilitation (PNF) is a tool designed to reduce the changes in respiratory function, the commitment of the respiratory muscles, and allows greater flexibility of the chest wall, reducing the rigidity of the rib cage. To evaluate the effects of respiratory pattern of Proprioceptive Neuromuscular Facilitation on the distribution of pulmonary ventilation, compartmental volumes of diaphragmatic mobility and functional capacity in patients with Parkinson's disease.

METHODS:

The study is a clinical trial randomized, in which participants to be elected for the study should present diagnosis of PD, staging of disease between II and III according to Hoehn and Yahr. Initially, the participants will undergo the collection of data on medical history, assessment of pulmonary function by spirometry and respiratory muscle strength measured by the manometer. Then will undergo evaluation of the breathing pattern and tricompartmental distribution of the volume of the chest wall by hemithorax by Plethysmography Optoelectronic; Quantify the mobility of the right diaphragm in total lung capacity for maneuver and during the current volume by ultrasonography. After the evaluation, participants will undergo intervention which will consist of three stages: first occur first session of the PNF later aerobic training for 30 minutes, ending with one PNF session.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with stage II and III between the Hoehn and Yahr classification;
* minimum score of 28 on the Mini Mental Examination for Parkinson.

Exclusion Criteria:

* individuals with rheumatologic or orthopedic diseases or deformities / abnormalities in the spine that compromise the respiratory mechanics;
* respiratory comorbidities;
* history of smoking;
* history of thoracic or abdominal surgery;
* clinical instability characterized by infections and / or hemodynamic defined as greater than 150 bpm heart rate or systolic blood pressure less than 90 mmHg;
* Not present exchange of the drug in the last 30 days.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
LUNG VOLUME | 1 MONTH
  BY OPTOELECTRONIC PLETHYSMOGRAPHY
WALKING DISTANCE, VO2, VCO2 | 1 MONTH
  SIX-MINUTE WALK TEST PLUS CÓRTEX

SECONDARY OUTCOMES:
DIAPHRAGM MOBILITY | 1 MONTH
  ULTRASOUND
DIAPHRAGM THICKNESS | 1 MONTH
  ULTRASOUND

OTHER OUTCOMES:
PRESSURE RESPIRATORY MAXIMAL | 1 MONTH
  BY MANOVACUOMETER

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Costa A, Bagoj E, Monaco M, Zabberoni S, De Rosa S, Mundi C, Caltagirone C, Carlesimo GA. Mini mental Parkinson test: standardization and normative data on an Italian sample. Neurol Sci. 2013 Oct;34(10):1797-803. doi: 10.1007/s10072-013-1342-8. Epub 2013 Mar 12. PMID 23479031
- [Background] Isella V, Mapelli C, Morielli N, De Gaspari D, Siri C, Pezzoli G, Antonini A, Poletti M, Bonuccelli U, Picchi L, Napolitano A, Vista M, Greco A, Appollonio IM. Validity and metric of MiniMental Parkinson and MiniMental State Examination in Parkinson's disease. Neurol Sci. 2013 Oct;34(10):1751-8. doi: 10.1007/s10072-013-1328-6. Epub 2013 Feb 20. PMID 23423464
- [Background] Carvalho A, Barbirato D, Araujo N, Martins JV, Cavalcanti JL, Santos TM, Coutinho ES, Laks J, Deslandes AC. Comparison of strength training, aerobic training, and additional physical therapy as supplementary treatments for Parkinson's disease: pilot study. Clin Interv Aging. 2015 Jan 7;10:183-91. doi: 10.2147/CIA.S68779. eCollection 2015. PMID 25609935
- [Background] Pereira CA, Sato T, Rodrigues SC. New reference values for forced spirometry in white adults in Brazil. J Bras Pneumol. 2007 Jul-Aug;33(4):397-406. doi: 10.1590/s1806-37132007000400008. English, Portuguese. PMID 17982531
- [Background] Aliverti A, Pedotti A. Opto-electronic plethysmography. Monaldi Arch Chest Dis. 2003 Jan-Mar;59(1):12-6. PMID 14533277
- [Background] Testa A, Soldati G, Giannuzzi R, Berardi S, Portale G, Gentiloni Silveri N. Ultrasound M-mode assessment of diaphragmatic kinetics by anterior transverse scanning in healthy subjects. Ultrasound Med Biol. 2011 Jan;37(1):44-52. doi: 10.1016/j.ultrasmedbio.2010.10.004. PMID 21144957
- [Background] Neder JA, Andreoni S, Lerario MC, Nery LE. Reference values for lung function tests. II. Maximal respiratory pressures and voluntary ventilation. Braz J Med Biol Res. 1999 Jun;32(6):719-27. doi: 10.1590/s0100-879x1999000600007. PMID 10412550
- [Background] MOORE, V. C. Spirometry: Step by step. Breathe, v. 8, n. 3, p. 233-240, 2012
- [Background] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402